CLINICAL TRIAL: NCT04213456
Title: Double Blind, Randomized, Placebo Controlled Pilot Study to Evaluate the Effect of Nutritional Supplementation on Physical Activity Performance of Young Soccer Players
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: NG Solutions Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RMC0888-18ctil
Record Dates: First submitted 2019-12-26; First posted 2019-12-30 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Nutritional Supplementation; Growth
Keywords: sport performance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional supplementation (Experimental): Powder added to water,high protein and multi vitamin and minerals
  Interventions: Dietary Supplement: Nutritional Sport Formula
- Placebo (Placebo Comparator): Low caloric formula (Powder added to water), without added vitamins and minerals.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nutritional Sport Formula — Powder added to water,high protein and multi vitamins and minerals
  Arms: Nutritional supplementation
Dietary Supplement: Placebo — Low caloric formula (Powder added to water), without added vitamins and minerals.
  Arms: Placebo

SUMMARY:
Research has clearly shown that lacking sufficient calories, macro- and micro-nutrients may impair an athlete's training adaptations, while athletes who consume a balanced diet that meets energy needs can enhance physiological training adaptations. Maintaining an energy and nutrient deficient diet during training may lead to loss of muscle mass, strength, and bone mineral density, in addition to an increased susceptibility to illness and injuries, disturbances in immune, endocrine and reproductive function, and an increased prevalence of overreaching and/or overtraining. In children and adolescent athletes, an insufficient diet may additionally result in impaired physical growth. Incorporating good dietary practices as part of a training program is one way to help optimize training adaptations and prevent overtraining.

Based on this, nutritional supplementation is an effective and safe approach for attaining the high nutritional requirements of adolescent athletes, to help them maintain healthy growth. Nutritional supplementation could also improve their body composition, sport performance and general health. The primary objective of the proposed study is to evaluate the effect of dietary supplement versus placebo on growth and physical activity performance in young athletes. A total of 50 young soccer players (25 in each group) will participate in this Double blind, randomized, placebo controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Young soccer players aged 8-15 years old

Exclusion Criteria:

* Diagnosis of GH Deficiency or treatment with GH
* Any known chronic disease or dysmorphic syndrome including: organic brain diseases, neurological disease, past or current malignancy, chronic cardiac, renal or pulmonary problems, gastrointestinal disease including malabsorption and bone dysplasia.

Ages: 8 Years to 15 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Height SDS (standard deviation score) | at 4 months
  Change in standard deviation score of participant's height between baseline and 4 months
10m sprint score | at 4 months
  Change in 10m sprint score between baseline and 4 months (test the speed and acceleration of the player)
20m sprint score | at 4 months
  Change in 20m sprint score between baseline and 4 months (test the speed and acceleration of the player)
Countermovement Jump (CMJ) score | at 4 months
  Change in Countermovement Jump (CMJ) score between baseline and 4 months (assess explosive strength of the lower extremity muscles)
Agility test score | at 4 months
  Change in Agility test score between baseline and 4 months(agility is the ability to change the direction of the body rapidly and is a result of a combination of strength, speed, balance and coordination)
The Yo-Yo Intermittent Recovery Test Level 1 (Yo-Yo IR1) score | at 4 months
  Change in the Yo-Yo IR1 score between baseline and 4 months (The Yo-Yo IR test measure the ability to recover from intense exercise)

SECONDARY OUTCOMES:
weight-SDS | at 4 months
  Change in standard deviation score of subject's weight between baseline and 4 months
BMI-SDS | at 4 months
  Change in standard deviation score of subject's BMI between baseline and 4 months

OTHER OUTCOMES:
Average daily caloric intake | at 4 months
Average daily macronutrients intake | at 4 months
Average daily micronutrients intake | at 4 months
Average weekly duration of physical activity | at 4 months
Average daily duration of sedentary activity | at 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Schnider Children's Medical Center, Petah Tikva, Israel